CLINICAL TRIAL: NCT07015281
Title: Dry Needling With Percutaneous Electrical Nerve Stimulation + Exercises Verus Therapeutic Execises in Patients With Non-specific Chronic Neck Pain
Brief Title: Dry Needling With Percutaneous Electrical Nerve Stimulation and Exercises for Non-specific Chronic Neck Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Responsible Party: Principal Investigator, Adelaida María Castro-Sánchez, PhD, Universidad de Almeria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP-0429-2023-C4-F3
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain
Keywords: exercise; quality of life; electrical stimulation; pain
MeSH Terms: conditions — Neck Pain; Motor Activity; Pain | interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation; Exercise Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling with Percutaneous Electrical Nerve Stimulation (PENS) and Therapeutic Exercises. (Experimental): Patients assigned to this group (n=50) will receive an intervention in which PENS will be applied for 30 minutes with low frequency parameters (2 Hz) and a pulse width of 120 μs. After 30 minutes of PENS in both groups, the needle will be removed and a compression will be applied for 90 seconds. Once the compression will carried out, the technique will be concluded. Patients will develop a session of PENS and a session with therapeutic exercise once a week.
  Interventions: Other: Therapeutic Exercise
- Therapeutic Exercise (Active Comparator): These participants (n=50) will engage in an exercise protocol with aerobic, isometric, resistence, strength, and stretching exercises. Participants will perform these exercises with a frequency of 3 times a week for 6 weeks, with each session lasting 30 minutes.
  Interventions: Other: Dry Needling with Percutaneous Electrical Nerve Stimulation (PENS) and Therapeutic Exercises.

INTERVENTIONS:
Other: Dry Needling with Percutaneous Electrical Nerve Stimulation (PENS) and Therapeutic Exercises. — Patients assigned to this group (n=50) will receive an intervention in which PENS will be applied for 30 minutes with low frequency parameters (2 Hz) and a pulse width of 120 μs. After 30 minutes of PENS in both groups, the needle will be removed and a compression will be applied for 90 seconds. Once the compression will carried out, the technique will be concluded. Patients will develop a session of PENS and a session with therapeutic exercise once a week.
  Other Names: Experimental
  Arms: Therapeutic Exercise
Other: Therapeutic Exercise — These participants (n=50) will engage in an exercise protocol with aerobic, isometric, resistence, strength, and stretching exercises. Participants will perform these exercises with a frequency of 3 times a week for 6 weeks, with each session lasting 30 minutes.
  Other Names: Active Comparator
  Arms: Dry Needling with Percutaneous Electrical Nerve Stimulation (PENS) and Therapeutic Exercises.

SUMMARY:
The aim of this study is to compare the effects of applying dry needling with percutaneous electrical nerve stimulation + exercises verus therapeutic execises in patients with non-specific chronic neck pain.

DETAILED DESCRIPTION:
Globally, neck pain is considered the fourth leading cause of years lived with disability. It is estimated that up to 70% of the world's population will experience neck pain at least once in their lifetime, and between 50% and 85% of cases will become chronic within a five-year period.

The point prevalence of neck pain in the adult population, aged 15-74 years, ranges from 5.9% to 38.7%. This prevalence has been observed to peak in the 50-74 age group. In 2017, the global age-standardized prevalence and incidence of neck pain were 3551.1 and 806.6 per 100,000 population, respectively.

Dry needling with percutaneous electrical nerve stimulation has positive short-term effects on pain intensity, pain-related disability, and mood in patients with chronic nonspecific neck pain, compared with no or minimal intervention. However, the long-term impact could not be assessed due to a lack of available studies. Furthermore, strong evidence has been found suggesting that dry needling with percutaneous electrical nerve stimulation may improve mental well-being and mood in patients with chronic neck pain, especially in those with pain induced by high levels of stress.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 30 and 65 years.
* A diagnosis of non-specific neck pain,
* Acceptance and signing of informed consent for voluntary participation in the research study.
* Not currently receiving physiotherapy.

Exclusion Criteria:

* Patients undergoing rehabilitative treatment for cervical pathologies.
* Patients with osteosynthesis material at the cervical level and/or cardiac, epileptic, or tumour-related complications.
* Patients who have undergone radiotherapy. in the last 6 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | At baseline, 6 weeks and 3 months (follow up).
  The neck disability index consists of 10 questions addressing functional activities such as personal care, lifting, reading, work, driving, sleeping, recreational, pain intensity, concentration and headache. Each item will be scored on a scale from 0 (no limitation). (severe limitation or inability to perform the activity). The total score will be calculated by summing the item scores, dividing by the maximum possible score of 50 (if all 10 questions are answered), and multiplying by 100 to generate a percentage. A score of 0% indicates full independence, while 100% represents complete dependence.

SECONDARY OUTCOMES:
Pain (Visual Analog Scale) | At baseline, 6 weeks and 3 months (follow up).
  Pain will be assessed with the Visual Analog Scale (VAS), which assesses the pain intensity and degree of relief experienced by the patient (scored of 0 = no pain; 10 = unbearable pain).
Quality of Life (SF-36 quality of life questionnaire). | At baseline, 6 weeks and 3 months (follow up).
  The SF-36 quality of life questionnaire assesses 8 domains including physical functioning, physical role, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Scores range from 0 to 100% (with higher scores indicating greater health), reflecting the individual's self-perceived health-related quality of life.
Quality of Sleep (Pittsburgh Quality of Sleep Questionnaire Index). | At baseline, 6 weeks and 3 months (follow up).
  The Pittsburgh Quality of Sleep Questionnaire Index (PSQI) will be used to study the quality of sleep. It comprises 24 items where the subjects respond to 19 of these items, and individual living in the same dwelling (or hospital room) responds to the remaining 5. Scores are obtained on each of 7 components of sleep quality: subjective quality, sleep latency, sleep duration, habitual sleep efficacy, sleep perturbations, use of hypnotic medication, and daily dysfunction. Using a four-point, Likert-type scale, respondents indicate how frequently they exhibit certain sleep behaviors (0 = "few," 1 = "sometimes," 2 = "often," and 3 = "almost always"). Scores on items belong to factors 2 and 5 (restoration after sleep and satisfaction with sleep) and are reversed before being tallied. Total scores can range from 0 to 84, with higher scores demoting more acute sleep problems.
Tampa scale for kinesiophobia. | At baseline, 6 weeks and 3 months (follow up).
  The 17-item Tampa scale for kinesiophobia assesses fear of movement or of injury or reinjury. Participants rate their beliefs regarding kinesiophobia on a 4-point Likert scale, ranging from "strongly disagree" to "strongly agree".
Pain Catastrophizing Scale. | At baseline, 6 weeks and 3 months (follow up).
  The Pain Catastrophizing Scale (PCS) is a self-assessment questionnaire to examine catastrophizing in clinical and nonclinical populations. Catastrophizing is commonly described as an exaggerated negative orientation toward noxious stimuli and plays an important role in experiencing and coping with pain. The PCS consists of 13 statements containing a number of thoughts and feelings one may experience when having pain. The items are divided into the categories of rumination, magnification and helplessness, with each item scored on a 5-point scale. The PCS consists of 13 statements containing several thoughts and feelings one may experience when having pain (scores 0-52).
Cervical Range of Motion (Pro Motion Capture. Werium). | At baseline, 6 weeks and 3 months (follow up).
  Cervical range of motion is assessed with the patient sitting comfortably on a chair, with both feet flat on the floor, hips and knees at 90º of flexion, and buttocks positioned against the back of the chair.
Spinal Isometric Strength (SIS). | At baseline, 6 weeks and 3 months (follow up).
  The investigators will measure the maximum isometric strength of the neck extensor muscles using a hand-held dynamometer (HHD). The patient will remain seated in a chair, with their feet flat on the floor, their hips and knees at 90º of flexion and the neck in the anatomical position, the patient will hold the HHD with both hands resting on their occiput, opposing the extension, and will be asked to perform a progressive isometric cervical extension for 3 seconds until reaching their maximum level of strength.
Neck Flexor Muscle Endurance Test (NFME). | At baseline, 6 weeks and 3 months (follow up).
  To measure the isometric endurance of the neck flexors, the investigators will place the patient in a supine position and ask him/her to perform a double chin tuck, which he/she must maintain throughout the test. While maintaining this position, he/she must flex his/her neck until his/her head is 2.5 cm off the table and maintain this position for as long as possible. The evaluator will time the duration of the test, which will be terminated if the patient loses the position for more than one second or asks to end due to fatigue or pain.
Treatment expectations. | At baseline, 6 weeks and 3 months (follow up).
  Questionnaire on treatment expectations and the patient's perception level.
Trigger points. | At baseline, 6 weeks and 3 months (follow up).
  Trigger oints will be measured in the following pairs of cervical muscles billaterally (right and left): occipitofrontalis, splenius capitis, sternocleidomastoid, anterior scalene, middele scalene, posterior scalene, upper trapezius, middle trapezius, lower trapezius, supraspinatus, infraspinatus, and multifidus level C6.

CONTACTS AND LOCATIONS:
Locations (1):
- Adelaida María Castro Sánchez, Almería, Almeria, Spain

IPD SHARING:
Plan to Share IPD: Yes
The study data will be available by email at adelaid@ual.es, provided that a reasonable request is made with justification for its scientific use and that citation is guaranteed.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning with the first article publication; ending 5 years following article publication.
Access Criteria: Data will be accessed via the contact email adelaid@ual.es, provided that its scientific use and citation of our protocol are guaranteed.

REFERENCES:
- [Background] Hernandez JVL, Calvo-Lobo C, Zugasti AM, Fernandez-Carnero J, Beltran Alacreu H. Effectiveness of Dry Needling with Percutaneous Electrical Nerve Stimulation of High Frequency Versus Low Frequency in Patients with Myofascial Neck Pain. Pain Physician. 2021 Mar;24(2):135-143. PMID 33740346
- [Background] Galasso A, Urits I, An D, Nguyen D, Borchart M, Yazdi C, Manchikanti L, Kaye RJ, Kaye AD, Mancuso KF, Viswanath O. A Comprehensive Review of the Treatment and Management of Myofascial Pain Syndrome. Curr Pain Headache Rep. 2020 Jun 27;24(8):43. doi: 10.1007/s11916-020-00877-5. PMID 32594264
- [Background] Chen IW, Liao YT, Tseng H, Lin HC, Chou LW. Pain, function and peritendinous effusion improvement after dry needling in patients with long head of biceps brachii tendinopathy: a single-blind randomized clinical trial. Ann Med. 2024 Dec;56(1):2391528. doi: 10.1080/07853890.2024.2391528. Epub 2024 Aug 14. PMID 39140690
- [Background] Moro MZ, de Oliveira Vidal EI, Pinheiro Modolo NS, Bono Fukushima F, Moreira de Barros GA. Dry needling, trigger point electroacupuncture and motor point electroacupuncture for the treatment of myofascial pain syndrome involving the trapezius: a randomised clinical trial. Acupunct Med. 2024 Feb;42(1):3-13. doi: 10.1177/09645284231207865. Epub 2023 Oct 31. PMID 37905789
- [Background] Leon-Hernandez JV, Martin-Pintado-Zugasti A, Frutos LG, Alguacil-Diego IM, de la Llave-Rincon AI, Fernandez-Carnero J. Immediate and short-term effects of the combination of dry needling and percutaneous TENS on post-needling soreness in patients with chronic myofascial neck pain. Braz J Phys Ther. 2016 Jul 11;20(5):422-431. doi: 10.1590/bjpt-rbf.2014.0176. PMID 27410163
- [Background] Baumann AN, Fiorentino A, Oleson CJ, Leland JM 3rd. The Impact of Dry Needling With Electrical Stimulation on Pain and Disability in Patients With Musculoskeletal Shoulder Pain: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. Cureus. 2023 Jul 5;15(7):e41404. doi: 10.7759/cureus.41404. eCollection 2023 Jul. PMID 37546088
- [Background] G A, Gupta AK, Kumar D, Mishra S, Yadav G, Singha Roy M, Prajapti L. Efficacy of Dry Needling Versus Transcutaneous Electrical Nerve Stimulation in Patients With Neck Pain Due to Myofascial Trigger Points: A Randomized Controlled Trial. Cureus. 2023 Mar 21;15(3):e36473. doi: 10.7759/cureus.36473. eCollection 2023 Mar. PMID 37090321
- [Background] Brennan K, Elifritz KM, Comire MM, Jupiter DC. Rate and maintenance of improvement of myofascial pain with dry needling alone vs. dry needling with intramuscular electrical stimulation: a randomized controlled trial. J Man Manip Ther. 2021 Aug;29(4):216-226. doi: 10.1080/10669817.2020.1824469. Epub 2020 Sep 29. PMID 32990529